CLINICAL TRIAL: NCT06387693
Title: Artificial Intelligence-assisted Diagnostics In Angina With No Obstructive Coronary Artery Disease
Brief Title: Artificial Intelligence in ANOCA
Acronym: (AI)NOCA
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: UMC Utrecht (Other)
Responsible Party: Principal Investigator, Tim P. van de Hoef, Principal Investigator, UMC Utrecht
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 24U-1359
Record Dates: First submitted 2024-04-03; First posted 2024-04-29 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2026-01

CONDITIONS: Angina, Stable
MeSH Terms: conditions — Angina, Stable | interventions — Electrocardiography, Ambulatory

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Single arm (Experimental): Intracoronary ECG and Holter ECG monitoring
  Interventions: Diagnostic Test: Holter monitoring, intracoronary ECG

INTERVENTIONS:
Diagnostic Test: Holter monitoring, intracoronary ECG — Holter monitoring device to track ECG abnormalities during spontaneous chest pain in the outpatient setting. Intracoronary ECG to evaluate perprocedural ECG responses

SUMMARY:
Angina pectoris is diagnosed in >180.000 people in the Netherlands each year. Diagnosis in angina pectoris focuses on epicardial coronary stenosis, the identification of which may lead to guideline-directed medical therapy or revascularization. However, no such stenosis is identified in 40-70% of patients. This condition, angina with no obstructed coronary artery (ANOCA), is more prevalent in women and is related to poor quality of life, high medical expenses, and a higher incidence of adverse events.

The origin of ANOCA can be evaluated during invasive coronary angiography by coronary function testing (CFT) to identify coronary vasomotor disorders. This relates to vasospasm of the coronary artery and microcirculation, or to impaired microvascular vasodilation. For the diagnosis of vasospasm, CFT needs to result in electrocardiographic signs of myocardial ischemia as part of the diagnostic criteria. This is a critical point in the diagnosis of vasospasm, as these signs can be subtle and can vary, and are therefore prone to misinterpretation. Apart from this caveat, the diagnosis approach therefore currently requires an invasive procedure for the diagnosis. This limits the broad application and hampers early identification and treatment of ANOCA.

During CFT, a coronary guide wire is routinely advanced in the coronary artery which also allows obtaining an intracoronary ECG by attaching a sterile alligator clamp to a standard electrocardiogram lead. This allows continuous recording of intracoronary ECG throughout CFT on the same monitor as the routine ECG. This technique can increase sensitivity for myocardial ischemia during CFT. Further, Holter ECG monitoring allows the identification of ischemic changes in the ECG in the outpatient setting. Evidence is lacking on the patterns of myocardial ischemia that occur during spontaneous angina pectoris symptoms in ANOCA patients, and on the sensitivity of Holter ECG for this purpose. Finally, the interpretation of ischemic patterns on ECG tracings can be cumbersome, especially when changes are subtle or change from beat to beat. The use of deep learning techniques allows to automate the interpretation of ECG traces and may improve the standardized diagnosis in ANOCA.

ELIGIBILITY:
Inclusion Criteria:

1. Clinical indication for comprehensive coronary function testing because of persisting chest discomfort at least 2 times per week despite current medical therapy.
2. Absence of obstructive coronary artery disease with an indication for revascularization, documented by means of recent coronary computed tomography angiography (CCTA) or invasive coronary angiography (with invasive coronary pressure measurements if clinically indicated).
3. Patient is willing and able to provide written informed consent.

Exclusion Criteria:

1. Absence of chest discomfort after initiation of medical therapy.
2. Language barrier preventing sufficient understanding and communication in Dutch.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250 (Estimated)
Dates: Start 2024-12-03 (Actual); Primary Completion 2028-08 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Prevalence of myocardial ischemia in patients with equivocal coronary function test results | During the procedure
  The prevalence of ischemic changes on the intracoronary ECG in patients with equivocal coronary function test results.
Diagnostic accuracy of perprocedural Holter ECG monitoring to diagnose coronary vasomotor disorders | During the procedure
  Accuracy of the Holter ECG to identify ischemic ECG changes compared with the standard 12-lead ECG during acetylcholine-provoked chest pain.
Diagnostic ccuracy of outpatient Holter monitoring for coronary vasomotor disorders | 7 days
  Diagnostic accuracy of outpatient Holter monitoring to diagnose vasomotor disorders using the coronary function test results as the reference standard

CONTACTS AND LOCATIONS:
Locations (1):
- UMC Utrecht, Utrecht, Netherlands

IPD SHARING:
Plan to Share IPD: Yes
IPD will be made available upon reasonable request.
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: A fully anonymized data set containing data from those patients who agreed with data sharing will be available upon reasonable request 12 months after finalization of the study.